CLINICAL TRIAL: NCT01576731
Title: Open Randomized Study Comparing Two Alternatives of Antiretroviral Therapy as Post-exposure Prophylaxis to HIV-1: Tenofovir + Emtricitabine + Lopinavir/Ritonavir Versus Tenofovir + Emtricitabine + Raltegravir
Brief Title: Study Comparing Two Alternatives of Antiretroviral Therapy as Post-exposure Prophylaxis to HIV-1: Tenofovir + Emtricitabine + Lopinavir/Ritonavir Versus Tenofovir + Emtricitabine + Raltegravir (RAL-PEP)
Acronym: RAL-PEP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Felipe Garcia, MD, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2011-003799-35
Record Dates: First submitted 2012-04-03; First posted 2012-04-12 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: HIV Infection
Keywords: HIV Infection; Postexposure prophylaxis
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir; Emtricitabine; Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tenofovir + emtricitabine + lopinavir/r (Active Comparator): Standard postexposure prophylaxis combination
  Interventions: Drug: Tenofovir, Emtricitabine, Lopinavir/r
- Tenofovir + Emtricitabine + Raltegravir (Experimental): new postexposure prophylaxis combination
  Interventions: Drug: Tenofovir, Emtricitabine, Raltegravir

INTERVENTIONS:
Drug: Tenofovir, Emtricitabine, Lopinavir/r — Combination drug
  Arms: Tenofovir + emtricitabine + lopinavir/r
Drug: Tenofovir, Emtricitabine, Raltegravir — Combination drug
  Arms: Tenofovir + Emtricitabine + Raltegravir

SUMMARY:
As a measure of secondary prophylaxis, and with the final objective of avoiding the infection, it has been suggested to use antiretroviral therapy. This is known as post-exposure prophylaxis (PEP).

Although there are different recommendations, almost every guideline recommend using 3 drugs as PEP both in USA and Europe.

Toxicity is one of the main limitations of PEP. Side effects during PEP are very usual, are attributed mainly to PI and are the main reasons for poor adherence or lost of follow-up.

A current standard regimen is AZT+3TC (Combivir®) or tenofovir+emtricitabine (Truvada®) plus the PI lopinavir/r. Toxicity associated with this regimens are high (31-85% of cases),with a high tolerability, a integrase inhibitor (raltegravir)could be an adequate drug for PEP.

ELIGIBILITY:
Inclusion Criteria:

* Potentially sexual exposition to HIV

Exclusion Criteria:

* Pregnancy
* Source case with antiretroviral resistances
* any treatment contraindicated with the drugs of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2012-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients dropping out before the 28 days of postexposure prophylaxis | 28 days
  Proportion of patients droppping out before the 28 days of postexposure prophylaxis considering death, lost to folow-up and stopping or changing treatment for any reason

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Garcia, PhD, Principal Investigator — Consultant senior
Locations (1):
- Hospital Clínic of Barcelona, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Leal L, Leon A, Torres B, Inciarte A, Lucero C, Mallolas J, Laguno M, Martinez-Rebollar M, Gonzalez-Cordon A, Manzardo C, Rojas J, Pich J, Arnaiz JA, Gatell JM, Garcia F; RALPEP Study Group. A randomized clinical trial comparing ritonavir-boosted lopinavir versus raltegravir each with tenofovir plus emtricitabine for post-exposure prophylaxis for HIV infection. J Antimicrob Chemother. 2016 Jul;71(7):1987-93. doi: 10.1093/jac/dkw049. Epub 2016 Mar 18. PMID 26994089